CLINICAL TRIAL: NCT02385903
Title: Randomized Controlled Trial on the Use of Flammacerium in Necrotic Arterial Wounds of the Lower Limb Versus Standard Treatment
Acronym: Flammacérium
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision of the Independent Review Committee
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Rangueil Hospital (Other); University Hospital, Caen (Other); Beziers Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8546
Record Dates: First submitted 2015-02-24; First posted 2015-03-11 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Ischemic Wound of the Lower Limb; Necrotic Arterial Wounds
Keywords: Flammacerium; Ischemic wound; Lower limb; Arteriopathy; Amputation; Dressing
MeSH Terms: interventions — cerous nitrate, sulfadiazine silver drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard dressing procedure (Other): One arm receive standard dressing procedure according to the wound
  Interventions: Other: Standard dressing procedure
- Flammacerium (Active Comparator): Necrosis covering with Flammacerium 3 mm thick each day during one week then one day on two.
  On each dressing, remove excess and add flammacerium. Not to remove crust forming until eliminating furrow appears.
  Cover Flammacerium by compress.
  Interventions: Other: Flammacerium

INTERVENTIONS:
Other: Flammacerium
  Arms: Flammacerium
Other: Standard dressing procedure
  Arms: Standard dressing procedure

SUMMARY:
Ischemia of an area may lead to a necrotic wound. In lower limb, it especially happens in diabetic or artheriopatic patients. It can lead to an amputation need. Revascularization procedure cannot be provide in all cases. Flammacerium, by a crust training and its anti-inflammatory effect, could stabilize necrosis extension, avoid bacterial contamination and then improve some incapacitating symptoms like odor or pain. This product may allow to delay amputation ruling for patients on who this procedure is unsafe. During 6 months, the investigators evaluate Flammacerium against standard dressing procedure in necrotic wound of the lower limb in patients where no revascularization can be provide. The investigators observed its effect on amputation need, symptoms as pain, infection, wound aspect evolution, wound size decrease.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic wound of the lower limb
* Minimum 50% necrosis
* Arteriopathy with ABI<0.7 or >1.3 with radiographic examinations
* No revascularisation procedure possible for any reasons
* No urgent amputation need
* Amputation considered in a short term
* Non life-threatened patients

Exclusion Criteria:

* Sulphonamide hypersensibility
* Propyleneglycols hypersensibility
* Enzyme glucose deshydrogenase deficiencies
* Others studies participation
* Tutorship or curatoship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-09; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Amputation rate | 6 months
  Level of amputation

SECONDARY OUTCOMES:
Infection rate | 6 months
Wound size | 6 months
Pain during dressing (VAS) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wound healing Department, Montpellier, France